CLINICAL TRIAL: NCT02085473
Title: A Phase 1 Study to Evaluate the Pharmacokinetics and Tolerability of a Single Subcutaneous Dose of Tralokinumab When Delivered as a 2 mL Injection at Different Flow Rates to Healthy Volunteers
Brief Title: A Study of Tralokinumab When Delivered Subcutaneously at Different Flow Rates to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D2210C00011
Record Dates: First submitted 2014-03-11; First posted 2014-03-12 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Asthma; Healthy Subjects or Volunteers
Keywords: Asthma; Healthy Subjects or Volunteers; Tralokinumab; CAT-354
MeSH Terms: conditions — Asthma | interventions — tralokinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Active Comparator): Participants received 300 milligram (mg) tralokinumab when delivered as a 2 milliliter (mL) subcutaneous injection at a flow rate of 'W' mL/min.
  Interventions: Biological: Tralokinumab 300 mg
- Cohort 2 (Experimental): Participants received 300 milligram (mg) tralokinumab when delivered as a 2 milliliter (mL) subcutaneous injection at a flow rate of 'X' mL/min.
  Interventions: Biological: Tralokinumab 300 mg
- Cohort 3 (Experimental): Participants received 300 milligram (mg) tralokinumab when delivered as a 2 milliliter (mL) subcutaneous injection at a flow rate of 'Y' mL/min.
  Interventions: Biological: Tralokinumab 300 mg
- Cohort 4 (Experimental): Participants received 300 milligram (mg) tralokinumab when delivered as a 2 milliliter (mL) subcutaneous injection at a flow rate of 'Z' mL/min.
  Interventions: Biological: Tralokinumab 300 mg

INTERVENTIONS:
Biological: Tralokinumab 300 mg — Participants will receive 300 milligram (mg) tralokinumab when delivered as a 2 milliliter (mL) subcutaneous injection at different flow rates.
  Other Names: CAT-354

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetics (PK) and tolerability of tralokinumab when delivered subcutaneously at different flow rates to healthy volunteers.

DETAILED DESCRIPTION:
This is a Phase 1, open-label, assessor-blind, parallel-group study to evaluate the PK and tolerability of a single subcutaneous dose of 300 milligram (mg) tralokinumab when delivered as a 2 milliliters (mL) injection at different flow rates to healthy adult volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy males and females ages 19-65 years
* Body mass index of 19.0-30.0 kilogram per meter square (kg/m^2)
* No clinically significant abnormality
* Vital signs, electrocardiogram (ECG), and laboratory parameters within normal range
* Negative alcohol and drug screens
* Females of childbearing potential who are sexually active with a nonsterilized male partner must use highly effective contraception
* Nonsterilized males who are sexually active with a female partner of childbearing potential must use highly effective contraception.

Key Exclusion Criteria:

* Concurrent enrollment in another clinical study where the subject is receiving an investigational product
* Receipt of any marketed or investigational biologic agent within 4 months or 5 half-lives prior to screening, whichever is longer
* Receipt of any investigational nonbiologic agent within 3 months or 5 half-lives prior to screening, whichever is longer
* Current use of regular pain-modifying, anti-depressant, anxiolytic, or hypnotic medication
* History of thrombocytopenia or bleeding disorder or use of anticoagulants
* History of any immunodeficiency disorder or use of immunosuppressive medication.
* History of a clinically significant infection
* History of cancer
* Positive Hepatitis B or C
* Positive HIV

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03-19 (Actual); Primary Completion 2014-07-10 (Actual); Study Completion 2014-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Cook, MD, Principal Investigator — Celerion
Locations (2):
- United States (2):
  - Celerion, Lincoln, Nebraska
  - Research Site, Lincoln, Nebraska

REFERENCES:
- [Background] Jain M, Doughty D, Clawson C, Li X, White N, Agoram B, van der Merwe R. Tralokinumab pharmacokinetics and tolerability when administered by different subcutaneous injection methods and rates . Int J Clin Pharmacol Ther. 2017 Jul;55(7):606-620. doi: 10.5414/CP203023. PMID 28590244
- See also: Redacted Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2689&filename=128095_Jain%20IJCPT_fully%20redacted%20protocol_23June17_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted between 19Mar2014 and 10Jul2014.
Pre-assignment Details: A total of 149 participants were screened for the study, out of which 60 participants were randomized and completed in the study.
Groups:
- Cohort 1: Participants received 300 milligram (mg) tralokinumab when delivered as a 2 milliliter (mL) subcutaneous injection at a flow rate of 6 mL/min.
- Cohort 2: Participants received 300 milligram (mg) tralokinumab when delivered as a 2 milliliter (mL) subcutaneous injection at a flow rate of 12 mL/min.
- Cohort 3: Participants received 300 milligram (mg) tralokinumab when delivered as a 2 milliliter (mL) subcutaneous injection at a flow rate of 2 mL/min.
- Cohort 4: Participants received 300 milligram (mg) tralokinumab when delivered as a 2 milliliter (mL) subcutaneous injection at a flow rate of 0.167 mL/min.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Started | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: As-treated population included all participants who were randomized and received any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.5 (9.5) | 39.7 (13.5) | 38.5 (14.1) | 38.4 (12.3) | 38.3 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 8 | 8 | 30
  Male | 8 | 8 | 7 | 7 | 30

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-Time Curve From Zero to Infinity (AUC [0-infinity])
Description: AUC (0 - infinity) = Area under the serum concentration versus time curve (AUC) from time zero to infinite time, obtained from AUC (0 - t) plus AUC (t - infinity). Units are day*micrograms per millilitres = day*mcg/mL.
Time Frame: Day 1 (pre-dose sample collected within 30 minutes prior to study drug administration), Days 2, 4, 6, 8, 10, 15, 22, 36, and 57 post-dose
Population: The Pharmacokinetic (PK) population included all participants in the as-treated population with at least one detectable tralokinumab serum concentration. Here "N" signifies participants who were evaluable for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*mcg/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 15 | 15 | 14 | 14
day*mcg/mL | 1426.47 (30.12) | 1243.28 (25.78) | 1251.63 (45.46) | 897.02 (39.13)

2. Primary Outcome: Maximum Observed Serum Concentration (Cmax)
Description: The Cmax is the maximum observed serum concentration of tralokinumab.
Time Frame: as for outcome 1
Population: The PK population included all participants in the as-treated population with at least one detectable tralokinumab serum concentration. Here "N" signifies participants who were evaluable for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 15 | 15 | 14 | 14
microgram per milliliter (mcg/mL) | 41.65 (28.20) | 34.07 (19.64) | 36.12 (35.69) | 27.04 (33.86)

3. Primary Outcome: Time to Maximum Concentration (Tmax)
Description: Tmax is defined as actual sampling time to reach maximum observed tralokinumab concentration.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: day
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 15 | 15 | 14 | 14
day | 8 [4 to 15] | 6 [4 to 10] | 8 [4 to 10] | 6 [4 to 10]

4. Primary Outcome: Area Under the Concentration-Time Curve From Zero to Last Measurable Concentration (AUC [0-t])
Description: AUC [0-t] is defined as area under the serum concentration-time curve from zero to last observed tralokinumab concentration.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*mcg/mL
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 15 | 15 | 14 | 14
day*mcg/mL | 1154.91 (25.92) | 998.08 (21.87) | 1013.98 (41.40) | 685.66 (35.85)

5. Primary Outcome: Terminal Elimination Half-life (t1/2)
Description: Terminal elimination half-life is the time measured for the serum concentration to decrease by one half. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 15 | 15 | 14 | 14
day | 21.62 (26.34) | 22.00 (24.11) | 21.91 (19.31) | 20.61 (20.74)

6. Primary Outcome: Apparent Systemic Clearance (CL/F) After Subcutaneous Dose
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after subcutaneous dose (apparent systemic clearance) is influenced by the fraction of the dose absorbed (bioavailability).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters per day (mL/day)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 15 | 15 | 14 | 14
milliliters per day (mL/day) | 210.31 (33.39) | 241.30 (29.16) | 239.69 (44.34) | 334.44 (355.50)

7. Primary Outcome: Apparent Terminal-Phase Volume of Distribution (Vz/F)
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters (mL)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 15 | 15 | 14 | 14
milliliters (mL) | 6559.99 (29.85) | 7657.96 (30.13) | 7577.56 (35.17) | 9944.14 (355.40)

8. Secondary Outcome: Local Injection-Site Pain and Injection-Site Pruritus
Description: Local injection-site pain and pruritus intensity was rated on 0 to 100 millimeter (mm) visual analogue scale (VAS) at various time points, where 0 = no pain/ no pruritus; 100 = most severe pain/ most severe pruritus. Injection site pruritus intensity was assessed by the blinded assessor. Higher the score indicated higher intensity of pain and pruritus. Local injection site pain and pruritus was assessed at below time-points: 1 and 6 minute (min) during investigational product administration (IPA); immediately post IPA, 10, 20, 30, and 60 min, 2, 4, 8, 24 and 72 hour (h) post IPA.
Time Frame: During the injection until 72 hours post-injection for injection site-pain and immediately after administration of injection until 72 hours for injection-site pruritus
Population: As-treated population included all participants who were randomized and received any study drug. Here, "N" signifies number of participants analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimole (mmol)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 15 | 15 | 15 | 15
millimole (mmol)
  Pain:1 min during IPA: number analyzed (Participants) | 0 | 0 | 0 | 15
  Pain:1 min during IPA |  |  |  | 6.7 (12.9)
  Pain:6 min during IPA: number analyzed (Participants) | 0 | 0 | 0 | 15
  Pain:6 min during IPA |  |  |  | 4.8 (5.9)
  Pain: Immediately Post IPA | 21.9 (20.9) | 41.0 (27.7) | 17.7 (15.5) | 5.1 (8.0)
  Pain:10 min Post IPA | 6.9 (13.9) | 7.1 (7.7) | 9.5 (16.3) | 1.3 (1.3)
  Pain:20 min Post IPA | 2.3 (5.0) | 3.7 (7.6) | 1.8 (2.6) | 1.2 (1.3)
  Pain:30 min Post IPA | 0.7 (1.0) | 1.3 (1.4) | 1.3 (2.2) | 1.2 (1.3)
  Pain:60 min Post IPA | 0.7 (1.0) | 1.1 (1.5) | 0.7 (1.0) | 1.2 (1.2)
  Pain:2h Post IPA | 0.3 (0.6) | 0.9 (1.3) | 0.8 (1.0) | 0.9 (1.6)
  Pain:4h Post IPA | 0.5 (0.7) | 0.9 (1.6) | 0.7 (0.9) | 1.0 (1.5)
  Pain:8h Post IPA | 0.5 (0.7) | 0.7 (1.4) | 0.5 (0.7) | 1.1 (1.6)
  Pain:24h Post IPA | 0.4 (0.6) | 0.7 (1.6) | 0.4 (0.6) | 0.9 (1.4)
  Pain:72h Post IPA | 0.6 (0.8) | 1.1 (1.7) | 0.5 (0.8) | 0.8 (1.2)
  Pruritus:Immediately Post IPA | 4.8 (7.5) | 15.1 (20.2) | 4.0 (5.6) | 6.9 (15.5)
  Pruritus:10 min Post IPA | 0.9 (0.9) | 3.1 (3.8) | 1.9 (2.3) | 4.1 (11.1)
  Pruritus:20 min Post IPA | 0.7 (0.8) | 1.9 (2.0) | 1.5 (1.5) | 2.5 (3.8)
  Pruritus:30 min Post IPA | 0.5 (0.7) | 1.1 (1.4) | 0.9 (1.3) | 1.8 (1.8)
  Pruritus:60 min Post IPA | 0.6 (0.8) | 1.0 (1.9) | 0.7 (1.0) | 1.3 (1.1)
  Pruritus:2h Post IPA | 0.4 (0.6) | 0.7 (1.3) | 0.7 (1.0) | 0.8 (1.3)
  Pruritus:4h Post IPA | 0.6 (0.7) | 0.8 (1.4) | 0.6 (0.7) | 0.9 (1.4)
  Pruritus:8h Post IPA | 0.4 (0.6) | 1.1 (1.8) | 0.7 (0.6) | 1.2 (2.0)
  Pruritus:24h Post IPA | 0.6 (0.7) | 0.6 (1.5) | 0.3 (0.6) | 0.7 (1.3)
  Pruritus:72h Post IPA | 0.5 (0.8) | 1.0 (1.4) | 0.6 (1.0) | 0.7 (1.0)

9. Secondary Outcome: Number of Participants Reporting Local Injection-Site Reactions
Description: The signs and/or symptoms of local injection-site reactions including erythema, hematoma or bleeding, local warmth, swelling, and/or rash occurring within 72 hours post-injection were assessed and recorded by a blinded assessor.
Time Frame: 0, 10, 20, 30 and 60 minutes, 2, 4, 8, 24 and 72 hours post-injection
Population: As-treated population included all participants who were randomized and received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants
  Erythema | 7 | 5 | 12 | 11
  Hematoma or bleeding | 2 | 1 | 3 | 5
  Local warmth | 0 | 0 | 0 | 0
  Swelling | 0 | 0 | 0 | 0
  Rash | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly and important medical event. Treatment-emergent were events between administration of study drug and up to Day 57 that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: From start of study drug administration up to Day 57
Population: As-treated population included all participants who were randomized and received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants
  TEAEs | 5 | 5 | 4 | 4
  TESAEs | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants Reporting Treatment-emergent Adverse Events Related to Physical Examination
Description: The treatment-emergent adverse events related to physical examination were reported as per investigator discretion. Treatment-emergent were the events between administration of study drug and up to Day 57 that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Day 1 to Day 57
Population: As-treated population included all participants who were randomized and received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants Reporting Treatment-emergent Adverse Events Related to Vital Signs
Description: Vital signs included systolic blood pressure, diastolic blood pressure, heart rate, respiratory rate and temperature. The treatment-emergent adverse events related to vital signs were reported as per investigator discretion. Treatment-emergent were the events between administration of study drug and up to Day 57 that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Day 1 to Day 57
Population: As-treated population included all participants who were randomized and received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants Reporting Treatment-emergent Adverse Events in Laboratory Parameters
Description: Laboratory parameters included hematology, serum chemistry and urinalysis. The treatment-emergent adverse events in laboratory parameters were reported as per investigator discretion. Treatment-emergent were the events between administration of study drug and up to Day 57 that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Day 1 to Day 57
Population: As-treated population included all participants who were randomized and received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants
  Hematology | 0 | 0 | 0 | 0
  Serum Chemistry | 0 | 0 | 0 | 0
  Urinalysis | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants Exhibiting Anti-Drug Antibodies for Tralokinumab at Any Visit
Description: Immunogenicity assessment included determination of anti-drug antibodies to tralokinumab (CAT-354) antibodies in serum samples.
Time Frame: Pre-dose on Day 1 and Day 57
Population: As-treated population included all participants who were randomized and received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Day 57
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 5/15 | 5/15 | 4/15 | 4/15
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=15) | Cohort 2 (N=15) | Cohort 3 (N=15) | Cohort 4 (N=15)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3) | 3 (3) | 3 (3)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.